CLINICAL TRIAL: NCT05879809
Title: Effect of Music Therapy in Depressive Symptoms of Mood Disorder: A Randomized Controlled Trial
Brief Title: Effect of Music Therapy in Depressive Symptoms of Mood Disorder（EMTDSMD）
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu Province Nanjing Brain Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 81725005-5
Record Dates: First submitted 2023-05-19; First posted 2023-05-30 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-04

CONDITIONS: Mood Disorder (Depressive Episodes)
MeSH Terms: conditions — Mood Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The clinical response of the MT (Experimental): To assess the efficacy of music therapy of MT group compared to control group in depressive symptoms.
  Interventions: Device: The mini apps named "SOUL GYM" on the Wechat
- The alterations of acoustic features in the MT (Experimental): To understand the possible biological mechanism underlying the efficacy of music therapy by analyzing alterations of acoustic features.
  Interventions: Device: The mini apps named "SOUL GYM" on the Wechat
- The alterations of neuroimaging features in the MT (Experimental): To investigate potential neurobiological mechanisms underlying the effectiveness of music therapy by analyzing alterations in neuroimaging features.
  Interventions: Device: The mini apps named "SOUL GYM" on the Wechat

INTERVENTIONS:
Device: The mini apps named "SOUL GYM" on the Wechat — Music Therapy can make peoples gradually relax via relaxing and soothing music, and regulate individual psychological emotions through the influence of music on individuals. The clinical symptoms will be evaluated before and after MT intervention.
  Arms: The clinical response of the MT
Device: The mini apps named "SOUL GYM" on the Wechat — Music Therapy can make peoples gradually relax via relaxing and soothing music, and regulate individual psychological emotions through the influence of music on individuals. The acoustic features will be evaluated before and after MT intervention.
  Arms: The alterations of acoustic features in the MT
Device: The mini apps named "SOUL GYM" on the Wechat — Music Therapy can make peoples gradually relax via relaxing and soothing music, and regulate individual psychological emotions through the influence of music on individuals. The neuroimaging features will be evaluated before and after MT intervention.
  Arms: The alterations of neuroimaging features in the MT

SUMMARY:
Depressive symptom is a common symptom that can be present in various psychiatric conditions, including depression and bipolar disorder. If left untreated, moderate to severe depressive symptoms can lead to serious health complications and are closely linked with suicide. Music therapy (MT)interventions have emerged as an important non-pharmacological approach to treating psychiatric and behavioral disorders, and have been observed to effectively alleviate depressive symptoms. Through its impact on the cerebral cortex, hypothalamus, and limbic system, music helps to regulate an individual's psychological state and can alleviate depressive symptoms.

This study utilized a randomized clinical trial design involving two groups: the MT group and the control group, both of which exhibited depressive symptoms. The MT group received MT in addition to routine clinical treatment, while the control group received only routine clinical treatment. The objective of this study was to demonstrate that MT is an effective intervention for alleviating depressive symptoms and to elucidate the neurobiological mechanisms of MT.

DETAILED DESCRIPTION:
This study is a double-blind randomized controlled trial aimed at evaluating the effectiveness of MT compared to a control group for major depressive disorder.

Participants will be randomly assigned in a 1:1 ratio to the MT group or control group. All participants will receive 12 sessions (3 sessions per week), each lasting 30 minutes, over a 4-week period. The MT group will receive music therapy during the first 4 weeks, while the control group will receive music therapy during the subsequent 4 weeks (weeks 5-8). Prior to the start of the study (baseline) and after the 4-week intervention, both groups will undergo symptom assessments and brain imaging (MRI) to collect data. The MT intervention consists of three stages, each with a specific focus: 1) physical and mental relaxation, which involves learning relaxation techniques from breathing to muscle relaxation; 2) nature imagination, which includes guided music imagery; and 3) internal self-exploration, which involves identifying positive experiences and potential resources for psychological intervention. The study aims to: 1) assess the clinical efficacy of MT in reducing depressive symptoms, and 2) examine possible biological mechanisms underlying the effectiveness of MT through multidimensional analysis of neuroimaging data and acoustic feature alterations.

ELIGIBILITY:
Inclusion Criteria:

* Between 13 and 35 years of age;
* Participants fulfill the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) diagnostic criteria for major depressive disorder (MDD) or bipolar disorder (BD). Participants are assessed by the Structured Clinical Interview for DSM-IV for Axis I Disorders (SCID-I, patients' age ≥18 years old), or the Schedule for Affective Disorders and Schizophrenia for School-Age Children-Present and Lifetime version (KSADS-PL, patients' age< 18 years old);
* A current depressive episode defined by HAMD≥7 and Young Mania Rating Scale (YMRS) <12;
* Participants receive a stable psychotropic medication regimen prior to randomization to the trial and are willing to remain on the stable regimen during the music treatment phase;
* Participants and 1 or 2 parents (patients' age< 18 years old) provide informed consent after the detailed description of the study.

Exclusion Criteria:

* • Prior music treatment or standard psychological therapy within 6 months prior to screening;

  * Comorbidity of other DSM-IV axis I disorders or personality disorders;
  * Judged clinically to be at serious suicidal risk;
  * Diabetes mellitus, hypertension, vascular and infectious diseases and other major medical comorbidities;
  * Unstable medical conditions, e.g., severe asthma;
  * Neurological disorders, e.g., history of head injury with loss of consciousness for ≥ five minutes, cerebrovascular diseases, brain tumors and neurodegenerative diseases;
  * Mental retardation or autism spectrum disorder;
  * Contraindications to MRI (e.g., severe claustrophobia, pacemakers, metal implants);
  * Current drug/alcohol abuse or dependence;
  * Pregnant or lactating female

Ages: 13 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in depressive symptoms assessed by the Patient Health Questionnaire-9 (PHQ-9; range: 0-27) at week 4. | Baseline and week 4
  The total scores of these questionnaires were interpreted as follows: normal (0-4), mild (5-9), moderate (10-14), and severe (15-27) depression.
Change from baseline in depressive symptoms assessed by Hamilton depression rating scale 17 items (HAMD-17) at week 4 | Baseline and week 4
  The HAMD-17 scale has 17 items. The total score ranges from 0-52, with higher score indicating more severe depressive symptoms. A total score of 0-7 is considered to be normal. Scores of 7 or higher indicate mild, moderate, severe, or very severe depression.
Change from baseline in the Clinical Global Impression-Severity scale (CGI-S) at week 4. | Baseline and week 4
  The CGI-S is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. A rating of 1 is considered normal, or with the least severe symptoms, a rating of 7 is extremely ill, or the worst symptoms.
Change from baseline in the Montgomery-Asberg Depression Rating Scale (MADRS) at week 4 | Baseline and week 4
  MADRS is a clinician-rated scale used to assess depressive symptom severity and detect changes due to antidepressant treatment. The scale consists of 10 items, each of which is rated from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms). The total score of MADRS ranges from 0 to 60, with higher score indicating more severe depression.
Change from baseline in anxiety symptoms assessed by the Generalized Anxiety Disorder-7 (GAD-7, range: 0-21) at week 4. | Baseline and week 4
  The total scores of these questionnaires were interpreted as follows: normal (0-4), mild (5-9), moderate (10-14), and severe (15-21) anxiety.
Change from baseline in insomnia symptoms assessed by the Insomnia Severity Index (ISI; range: 0-28) at week 4. | Baseline and week 4
  The total scores of these questionnaires were interpreted as follows: normal (0-7), mild (8-14), moderate (15-21), and severe (22-28) insomnia.
Change from baseline in perceived stress assessed by the Perceived Stress Scale-14 (PSS-14; range: 0-56) at week 4 | Baseline and week 4
  The total scores of these questionnaires were interpreted as follows: normal (0-28), moderate (29-42), severe (43-56).
Change from baseline in the amplitude of low-frequency fluctuation (ALFF) values measured by resting-state functional magnetic resonance imaging (fMRI) at week 4 | Baseline and week 4
  Participants will undergo fMRI scans prior to beginning music treatment (baseline) and after completing music treatment (week 4). ALFF is a fMRI indicator that reflects the spontaneous neural activity. After data acquisition, whole-brain voxel-wise analysis of ALFF values will be performed to detect the change from baseline in brain functional activity at baseline and week 4.

IPD SHARING:
Plan to Share IPD: Undecided